CLINICAL TRIAL: NCT02265809
Title: Adaptive Study of IL-2 Dose Frequency on Regulatory T Cells in Type 1 Diabetes (DILfrequency)
Brief Title: Adaptive Study of IL-2 Dose Frequency on Regulatory T Cells in Type 1 Diabetes
Acronym: DILfrequency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Sir Jules Thorn Charitable Trust (Unknown); Juvenile Diabetes Research Foundation (Other); Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr Frank Waldron-Lynch, Academic Consultant Endocrinologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DILfrequency
Record Dates: First submitted 2014-10-08; First posted 2014-10-16 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes
Keywords: Interleukin 2; Type 1 diabetes; T regulatory cells; Adaptive trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aldesleukin (Experimental): Aldesleukin will be administered subcutaneously at varying doses and frequencies for a period of up to 98 days from first administration depending on the treatment assignment. The maximum dose allowed is 0.6 X 10^6 IU/m2.
  Interventions: Drug: Aldesleukin

INTERVENTIONS:
Drug: Aldesleukin
  Other Names: Proleukin; IL-2

SUMMARY:
Type 1 diabetes (T1D) is the most common severe autoimmune disease worldwide and is caused by the body's immune destruction of its own insulin producing pancreatic beta cells leading to insulin deficiency and development of elevated blood sugars. Currently, medical management of T1D focuses on intensive insulin replacement therapy to limit complications (retinopathy, nephropathy, neuropathy); nevertheless clinical outcomes remain suboptimal. There are intensive efforts to design novel immunotherapies that can arrest the autoimmune process and thereby preserve residual insulin production leading to fewer complications and better clinical outcomes.

Genetics are in part the cause of T1D and the majority of genes contributing to T1D produce proteins involved in immune regulation (called "tolerance"). A key player in immune tolerance is a molecule called interleukin-2 (IL-2) which enhances the ability of cells called T regulatory (Treg) cells to suppress the destruction the insulin producing beta cells. Aldesleukin is a human recombinant IL-2 product produced by recombinant DNA technology using a genetically engineered E. coli strain expressing an analogue of the human IL-2 gene. There is substantial data to suggest that ultra-low doses (ULD) of IL-2 (aldesleukin) can arrest the autoimmune mediated destruction of pancreatic beta cells by the induction of functional Treg cells.

The former study "Adaptive study of IL-2 dose on regulatory T cells in type 1 diabetes" (DILT1D) (NCT 01827735) was a single dose mechanistic study designed to establish the doses of IL-2 (aldesleukin) required to induce a minimal Treg increase (0.1 fold from baseline) or to induce a slightly larger Treg increase (0.2 fold from baseline) (maximal increase). Following on from the DILT1D study, the goal of the DILfrequency study is to use an adaptive design to determine the optimal dose and frequency of ULD IL-2 (aldesleukin) to maximize Treg function by frequently injecting ultra-low doses of IL-2 (aldesleukin). The responsiveness of each T1D participant to a particular frequency of IL-2 (aldesleukin) administration informs the frequency of dosing given to the next patient. This strategy focuses on improving the function of regulatory T cells that are exquisitely sensitive to IL-2 (aldesleukin).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* 18-70 years of age
* Duration of diabetes less than 60 months from diagnosis
* Written informed consent to participate

Exclusion Criteria:

* Hypersensitivity to aldesleukin or any of the excipients
* History of severe cardiac disease
* History of malignancy within the past 5 years (with the exception of localized carcinoma of the skin that had been resected for cure or cervical carcinoma in situ)
* History or concurrent use of immunosuppressive agents or steroids
* History of unstable diabetes with recurrent hypoglycaemia
* History of live vaccination two weeks prior to first treatment
* Active autoimmune hyper or hypothyroidism
* Active clinical infection
* Major pre-existing organ dysfunction or previous organ allograft
* Females who are pregnant, lactating or intend to get pregnant during the study
* Males who intend to father a pregnancy during the study
* Donation of more than 500 ml of blood within 2 months prior to aldesleukin administration
* Participation in a previous therapeutic clinical trial within 2 months prior to aldesleukin administration
* Abnormal ECG
* Abnormal full blood count, chronic renal failure (Stage 3,4,5) and/or evidence of severely impaired liver function (ALT/AST > 3xULN at screening; alkaline phosphatase and bilirubin 2xULN at screening (isolated bilirubin >2xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%))

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline of CD4 T regulatory cells, CD4 T effector cells and CD25 expression on T regulatory cells during treatment with ultra low dose IL-2 | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Fluorescence-activated cell sorting

SECONDARY OUTCOMES:
T regulatory cell number, phenotype and proliferation | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by fluorescence-activated cell sorting
T effector cell number, phenotype and proliferation | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by fluorescence-activated cell sorting
Natural Killer cell number, phenotype and proliferation | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by fluorescence-activated cell sorting
B lymphocyte cell number, phenotype and proliferation | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by fluorescence-activated cell sorting
T cell and Natural killer cell intracellular signalling | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by fluorescence-activated cell sorting
Full blood count | Visits 1-12 (between day -30 and day -1 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by automatic analyser
Blood levels of IL-2, IL-6, IL-10, TNF-alpha, soluble CD25, IP-10, soluble rIL-6, and CRP | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by enzyme-linked immunosorbent assay
Change in metabolic control | Visits 1-12 (between day -30 and day -1 up to a maximum of approximately day 98 depending on treatment assignment)
  Blood glucose, HbA1c, C-peptide, insulin use and autoantibody status
Safety and tolerability | Visits 1-12 (between day -30 and day -1 up to a maximum of approximately day 98 depending on treatment assignment)
  Assessed by clinical history, physical examination, temperature, blood pressure, heart rate, 12-Lead electrocardiogram (ECGs), clinical laboratory tests, and adverse event recording

OTHER OUTCOMES:
Genotype of T1D associated loci | Visit 1 (between day -30 and day -1)
  Measured by immunochip
Gene expression analysis of purified lymphocyte subsets and peripheral blood mononucleated cells | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by RNA sequencing
IL-2 sensitivity of T regulatory, T effector and NK subsets | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by fluorescence-activated cell sorting
Treg suppression and T effector proliferation assays | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by radioactive thymidine assay and/or fluorescence-activated cell sorting
Antigen specific T cell assays | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured fluorescence-activated cell sorting and/or Enzyme-Linked ImmunoSpot (ELISPOT) assay
Sysmex® analysis of whole blood | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by automatic analyser
Epigenetic analysis of analysis of purified lymphocyte subsets and peripheral blood | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by Bisulphite sequencing of DNA
Serum/plasma level of cytokines, soluble receptors and inflammatory markers | Visits 2-12 (day 0 up to a maximum of approximately day 98 depending on treatment assignment)
  Measured by enzyme-linked immunosorbent assay
Serum/plasma and cellular metabolites | Visits 1-12 (between day -30 and day -1 up to a maximum of approximately day 98 depending on treatment assignment)
  Mass spectrometry
Recruitment analysis | Visit 1 (between day -30 and day -1)
  Analysis of DILfrequency recruitment database

CONTACTS AND LOCATIONS:
Overall Officials: Frank Waldron-Lynch, MB BChir PhD, Principal Investigator — University of Cambridge; Kevin M O'Shaughnessy, BM BCh DPhil, Study Chair — University of Cambridge
Locations (1):
- Wellcome Trust Clinical Research Facility, Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Waldron-Lynch F, Kareclas P, Irons K, Walker NM, Mander A, Wicker LS, Todd JA, Bond S. Rationale and study design of the Adaptive study of IL-2 dose on regulatory T cells in type 1 diabetes (DILT1D): a non-randomised, open label, adaptive dose finding trial. BMJ Open. 2014 Jun 4;4(6):e005559. doi: 10.1136/bmjopen-2014-005559. PMID 24898091
- [Background] Truman LA, Pekalski ML, Kareclas P, Evangelou M, Walker NM, Howlett J, Mander AP, Kennet J, Wicker LS, Bond S, Todd JA, Waldron-Lynch F. Protocol of the adaptive study of IL-2 dose frequency on regulatory T cells in type 1 diabetes (DILfrequency): a mechanistic, non-randomised, repeat dose, open-label, response-adaptive study. BMJ Open. 2015 Dec 8;5(12):e009799. doi: 10.1136/bmjopen-2015-009799. PMID 26646829
- [Derived] Zhang JY, Whalley JP, Knight JC, Wicker LS, Todd JA, Ferreira RC. SARS-CoV-2 infection induces a long-lived pro-inflammatory transcriptional profile. Genome Med. 2023 Sep 12;15(1):69. doi: 10.1186/s13073-023-01227-x. PMID 37700317
- [Derived] Seelig E, Howlett J, Porter L, Truman L, Heywood J, Kennet J, Arbon EL, Anselmiova K, Walker NM, Atkar R, Pekalski ML, Rytina E, Evans M, Wicker LS, Todd JA, Mander AP, Bond S, Waldron-Lynch F. The DILfrequency study is an adaptive trial to identify optimal IL-2 dosing in patients with type 1 diabetes. JCI Insight. 2018 Oct 4;3(19):e99306. doi: 10.1172/jci.insight.99306. PMID 30282826
- See also: Facebook page — https://www.facebook.com/ClinicalTrialsType1Diabetes
- See also: Twitter page — https://twitter.com/t1diabetestrial
- See also: Pinterest page — http://www.pinterest.com/t1diabetestrial/